CLINICAL TRIAL: NCT03131375
Title: Dexmedetomidine Reduces Emergence Delirium in Children Undergoing Tonsillectomy With Propofol Anesthesia: a Prospective, Randomized, Double-blind, Single-center Study.
Brief Title: Dexmedetomidine Reduces Emergence Delirium in Children Undergoing Tonsillectomy With Propofol Anesthesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Athens General Children's Hospital "Pan. & Aglaia Kyriakou" (Other)
Responsible Party: Principal Investigator, Adelais Tsiotou, Consultant of the Anesthesiology Dept, MD, PhD, Athens General Children's Hospital "Pan. & Aglaia Kyriakou"
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Dexmedetomidine.1.2017
Record Dates: First submitted 2017-04-20; First posted 2017-04-27 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Emergence Delirium; Extubation Time; Heart Rate; Postoperative Analgesia; Blood Pressure
Keywords: dexmedetomidine; emergence delirium; anesthesia; propofol; children
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Adrenergic alpha-2 Receptor Agonists; Saline Solution; Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): In Group A: Anesthesia induction drugs: propofol , fentanyl , rocuronium iv. After induction, Group A receives a 50 ml NS infusion containing the drug Dexmedetomidine 1 mcg kg-1 slowly. Anesthesia maintainance drugs: propofol and remifentanil. Reversal of neuromuscular block drugs: Sugammadex according to TOF measurements. Postoperative analgesia drugs: nalbuphine 0.16 mg kg-1 . Monitoring devices: ECG, NIBP , ETCO2, SpO2, Bispectral index, Train of four ratio.
  Interventions: Drug: Dexmedetomidine; Device: Bispectral index; Device: Train of four ratio
- Group B (Placebo Comparator): In Group B: Anesthesia induction drugs: propofol , fentanyl , rocuronium iv. After induction, Group B receives a volume matched normal saline infusion slowly. Anesthesia maintainance drugs: propofol and remifentanil. Reversal of neuromuscular block drugs: Sugammadex according to TOF measurements. Postoperative analgesia drugs: nalbuphine 0.2 mg kg-1 . Monitoring devices: ECG, NIBP , ETCO2, SpO2, Bispectral index, Train of four ratio.
  Interventions: Drug: Normal saline; Device: Bispectral index; Device: Train of four ratio

INTERVENTIONS:
Drug: Dexmedetomidine — Group A and B: Anesthesia induction drugs:propofol, fentanyl, rocuronium . After induction of anesthesia: Group A receives a 50 ml NS infusion containing 1 mcg kg-1 Dexmedetomidine drug Group A and B: Atropine as an antisialagogue, dexamethasone, ondasetrone for the prevention of postoperative nausea and vomiting. Anesthesia maintainance: propofol, remifentanil and oxygen in air. End of surgery, the infusion of propofol and remifentanil stop and sugammadex for reversal of neuromuscular block is given. Postoperative analgesia by nalbuphine 0.2 mg kg-1 given before the end of surgery in Group B, and 0.16 mg kg-1 in Group A. Monitoring: ECG, NIBP, ETCO2, SpO2, Bispectral index , Train of four ratio.
  Other Names: alpha-2 agonist
  Arms: Group A
Drug: Normal saline — Group A and B: Anesthesia induction drugs:propofol, fentanyl, rocuronium . After induction of anesthesia: Group B receives a volume matched Normal saline infusion. Group A and B: Atropine as an antisialagogue, dexamethasone, ondasetrone for the prevention of postoperative nausea and vomiting. Anesthesia maintainance: propofol, remifentanil and oxygen in air. End of surgery, the infusion of propofol and remifentanil stop and sugammadex for reversal of neuromuscular block is given. Postoperative analgesia by nalbuphine 0.2 mg kg-1 given before the end of surgery in Group B. Monitoring: ECG, NIBP, ETCO2, SpO2, Bispectral index, Train of four ratio.
  Other Names: placebo
  Arms: Group B
Device: Bispectral index — Group A and B: Monitoring depth of anesthesia by BIS device and adjusting propofol infusion according to measurements, aiming to BIS values: 40-60
  Other Names: BIS
Device: Train of four ratio — Group A and B: Monitoring recovery of neuromuscular function with TOF-Watch device, to ensure TOFR equals or greater than 90% at the end of the procedure
  Other Names: TOF-Watch

SUMMARY:
Dexmedetomidine (DEX) is safe and effective in reducing ED following sevoflurane anesthesia. The investigators intend to study the efficacy of DEX in reducing ED in children undergoing tonsillectomy with and without adenoidectomy using total intravenous anesthesia (TIVA) with propofol .

ELIGIBILITY:
Inclusion Criteria:

* Children
* ASA I or II
* tonsillectomy with or without adenoidectomy

Exclusion Criteria:

* Allergy to dexmedetomidine
* Allergy to anesthetic drugs
* History of neurological disease
* History of neuromuscular disease
* History of renal disease
* History of hepatic disease
* craniofacial anomalies
* History of cardiac disease
* History of respiratory disease

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Emergence delirium in PACU | up to 30 min
  Presence or absence of Emergence delirium with and without dexmedetomidine assessed by Watcha scale

SECONDARY OUTCOMES:
Emergence delirium severity, assessed in PACU | up to 30 min
  Watcha score
Extubation time | up to15 min
  time interval between discontinuation of anesthetics and extubation
Heart rate | up to 45 min
  monitored intraoperatively ECG
Blood pressure | up to 45 min
  monitored intraoperatively NIBP

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Kalliardou, Consultant, Study Director — Director of the Anesthesiology Dept.
Locations (1):
- Childrens Hospital P. and A. Kyriakou Anesthesiology Department, Athens, Greece

IPD SHARING:
Plan to Share IPD: No